CLINICAL TRIAL: NCT02667730
Title: Correlation Between Acute Analgesia and Long-Term Function Following Ankle
Brief Title: Correlation Between Acute Analgesia and Long-Term Function Following Ankle Injuries
Acronym: CALF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Canadian Department of National Defence (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-12-126-004-0001
Record Dates: First submitted 2015-07-09; First posted 2016-01-29 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Ligament Injury
MeSH Terms: interventions — Acetaminophen; Naproxen; Celecoxib

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Patients are aware of their allocation. The treating physiotherapists will not be aware of allocation and patients are asked to not discuss their medication (allocation) with physiotherapists
Oversight: Data Monitoring Committee: No

ARMS (4):
- Physiotherapy only (Placebo Comparator): This group will receive non-pharmacological advice and physiotherapy only
  Interventions: Other: physiotherapy only
- Acetaminophen + physiotherapy (Experimental): This group will receive acetaminophen 500mg 4 times daily for 7 days in addition to standardized physiotherapy
  Interventions: Drug: Acetaminophen; Other: physiotherapy only
- Naproxen + physiotherapy (Experimental): This group will receive naproxen 500mg twice daily for 7 days in addition to standardized physiotherapy
  Interventions: Drug: Naproxen; Other: physiotherapy only
- Celecoxib + physiotherapy (Experimental): This group will receive celecoxib 100mg twice daily for 7 days in addition to standardized physiotherapy
  Interventions: Drug: Celecoxib; Other: physiotherapy only

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 500 mg four times daily for 7 days
  Other Names: tylenol
  Arms: Acetaminophen + physiotherapy
Drug: Naproxen — naproxen 500mg twice daily for 7 days
  Arms: Naproxen + physiotherapy
Drug: Celecoxib — celecoxib 100mg twice daily
  Other Names: celebrex
  Arms: Celecoxib + physiotherapy
Other: physiotherapy only — physiotherapy only (no drug)

SUMMARY:
In this 4-arm pragmatic randomized control trial, the investigators hope to decipher whether the use of non-opioid analgesics (naproxen, celecoxib, acetaminophen) in addition to standardized physiotherapy during the acute phase of grade I-II ankle injuries will result in functional differences compared to standardized physiotherapy alone

DETAILED DESCRIPTION:
Background Ankle sprains occur frequently in the Canadian Armed Forces (CAF) population and account for a significant proportion of lost work time. Equally significant is the use of analgesics (NSAID or non-NSAID) (NSAID = non steroidal anti-inflammatory drug) in the CAF population. Existing literature suggests that the rate and extent of soft tissue healing may be adversely affected by use of some analgesics, particularly non-steroidal anti-inflammatory agents (NSAIDs), when these are used immediately following joint injury. There have been two postulated mechanisms for this observation: the first being that inflammatory markers are required in the regeneration process; the second is that the diminished pain level as a result of analgesic use encourages overuse of the injured tissue. Unfortunately, the science is far from conclusive, since much of it is derived based on isolated exercises, conducted in experimental settings, in older populations, or extrapolated from biomarkers that have not been validated for clinical relevance. While there is no current standard of practice regarding the use of pain relievers following ankle injury, this practice continues to be widespread in the CAF.

Goal The proposed study aims to clarify whether three commonly used non-opioid pain relievers provide additional benefit or delay improvement in ankle function following mild ankle sprains, when compared to standardized physiotherapy treatment alone. The three agents investigated will be 1) the non-steroid anti-inflammatory drug naproxen, 2) the selective anti-inflammatory celecoxib, and 3) the centrally-acting analgesic acetaminophen.

Methods Patients presenting to the health clinic at Garrison Petawawa with acute ankle injuries will be screened for study eligibility. All individuals who elect to participate in this study will be referred for standardized physiotherapy treatment, which will be administered according to study protocol. Participants will also be randomized to one of four analgesic treatment groups (i.e., naproxen, celecoxib, acetaminophen, or non-pharmacological measures only), with stratification for grade of ankle injury. Physiotherapists who are blinded to analgesic treatment allocation will evaluate participants' ankle function at 72 hours, 2 weeks, 3 months and 1 year post-injury, using previously validated tests. Pharmacists will assess response to drug therapy, side effects, and use of rescue medications at day 7 following enrollment. Occurrence of repeat ankle injuries and health resource consumption (i.e., specialist visits and diagnostic imaging) will also be assessed for the year following index injury.

Risks This study is intended to be low risk to participants as it is designed to closely mirror existing practices for such injuries. All medications used in this study are indicated for soft tissue injuries and their respective dosages/frequencies/durations aligned with manufacturer recommendations. The physiotherapy intervention was developed by Dr. Eric Robitaille. It has been used in previous studies and is currently in use in the CAF. The investigators do not expect the risk of injury to be higher than that associated with existing practices for ankle injuries.

Benefits Participants are expected to benefit from the direct application of a standardized physiotherapy treatment protocol for overall management of their condition as well as the pain relief from the analgesic options. The results of this study are expected to generate new information that can be readily applied to patient care, specifically in treating a frequently-occurring soft tissue injury in the CAF population.

ELIGIBILITY:
Inclusion Criteria:

* Acquired acute ankle injury (injured less than 48 hours ago);
* Clinical diagnosis of a Grade I or II ankle sprain
* Is eligible to receive comprehensive medical care from Garrison Petawawa

Exclusion Criteria:

* Diagnosis of ankle fracture or ligament rupture
* Has planned release from the Canadian Armed Forces within one year;
* Documented restrictions on military duties
* Has known intolerance or documented adverse reaction to acetaminophen or naproxen or celecoxib
* Documented history of liver or kidney problems
* pregnant or breastfeeding

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Ankle Function on FAAM | 3 months
  Foot and Ankle Abilities Measure

SECONDARY OUTCOMES:
Pain on visual analogue scale (VAS) | 3 months
  visual analogue scale
Mobility on Wall Lunge | 3 months
  wall lunge test for ankle mobility
Laxity on anterior drawer test | 3 months
  test for laxity
Proprioception on SEBT | 3 months
  star excursion balance test
composite of health resource consumption | 1 year
  # of orthopedic specialist consults, diagnostics, patient encounters for MSK reasons, # of days off work

CONTACTS AND LOCATIONS:
Overall Officials: Koren Lui, BScPHM, Principal Investigator — Canadian Forces Health Services Group
Locations (1):
- 2 Fd Amb medical clinic, Petawawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No